CLINICAL TRIAL: NCT05740007
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Adaptive Study to Evaluate the Efficacy, Safety, and Tolerability of 2 Dose Levels of IW-3300 Administered Rectally for 12 Weeks to Treat Bladder Pain in Subjects With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: A Phase 2 Study of IW-3300 for the Treatment of Bladder Pain in Subjects With Interstitial Cystitis/Bladder Pain Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C3300-201
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IW-3300 100 µg (Experimental): IW-3300 at 100 µg rectal foam administered daily for 12 weeks
  Interventions: Drug: IW-3300 rectal foam
- IW-3300 300 µg (Experimental): IW-3300 at 300 µg rectal foam administered daily for 12 weeks
  Interventions: Drug: IW-3300 rectal foam
- Placebo (Placebo Comparator): Placebo rectal foam administered daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-3300 rectal foam — IW-3300 rectal foam administered daily for 12 weeks
  Arms: IW-3300 100 µg; IW-3300 300 µg
Drug: Placebo — Placebo rectal foam administered daily for 12 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is to assess whether IW-3300 is safe and works for the treatment of interstitial cystitis/bladder pain syndrome (IC/BPS). The main question the study aims to answer is whether IW-3300 helps bladder pain and other symptoms (for example, bladder burning, pressure and discomfort). Subjects will be assigned to receive either the study drug or placebo by chance.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, placebo-controlled, parallel-assignment, 12-week, adaptive design study to evaluate the efficacy, safety, and tolerability of IW-3300 in subjects with IC/BPS. Subjects will be randomized 1:1:1 to IW-3300 100 µg, IW-3300 300 µg, or matching placebo administered as a rectal foam. The study has 4 periods, which are the screening (up to 30 days), pretreatment (up to 21 days), study treatment (12 weeks), and follow-up periods (2 weeks) which consists of 7 onsite study visits and 1 follow-up phone call. Subjects will administer the study drug at home for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IC/BPS by a urologist or other clinician specializing in IC/BPS
* Chronic bladder pain associated with filling the bladder over the past 6 months
* Compliant with eDiary completion and meets weekly average daily score for bladder pain at its worst during the pretreatment period
* Has at least 1 of the following urinary symptoms over the past 6 months: nocturia ≥2 voids/night, daytime frequency >8×day, urgency
* Body mass index (BMI) ≤40 kg/m2
* Willing to use a rectally administered product once daily for 12 weeks

Exclusion Criteria:

* Male subject has history of bacterial prostatitis or benign prostatic hyperplasia with active symptoms that are difficult to distinguish from IC/BPS
* Has a condition that can be a contraindication to using a rectal foam
* Has cancer under active treatment or a history of uterine, cervical, pelvic, colorectal, ovarian, or vaginal cancer
* Has a history of benign or malignant bladder tumors
* Has an active urinary tract infection or had ≥2 UTIs within the past 90 days
* Has an uncontrolled major psychiatric condition or has made a suicide attempt during the past 2 years
* Has a malabsorption syndrome
* Had surgery in the pelvic or abdominal region within the past 90 days or is planning pelvic or abdominal region surgical procedures before the end of the study
* Has received a cystoscopy with or without hydrodistension for diagnostic purposes (ie, not for pain relief) within the past 30 days or a cystoscopy with therapeutic hydrodistension (ie, for pain relief) within the past 90 days or is planning a cystoscopy for any reason before the end of the study
* Has history of pelvic irradiation or radiation cystitis, or drug-induced cystitis.
* Has a recent history of drug or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline (CFB) in weekly average of daily bladder pain (which can include sensations like burning, pressure, and/or discomfort) at its worst at Week 12 | Baseline, Week 12
  Subject assessment of bladder pain at its worst will be reported via a daily electronic Diary (eDiary)

SECONDARY OUTCOMES:
CFB in weekly average of a burning sensation in the bladder at its worst at Week 12 | Baseline, Week 12
  Subject assessment of bladder burning sensation at its worst will be reported via an eDiary
CFB in weekly average of a pressure sensation in the bladder at its worst at Week 12 | Baseline, Week 12
  Subject assessment of bladder pressure sensation at its worst will be reported via an eDiary
CFB in weekly average of discomfort in the bladder at its worst at Week 12 | Baseline, Week 12
  Subject assessment of discomfort in the bladder at its worst will be reported via an eDiary
CFB in Genitourinary Pain Index (GUPI) Pain subscale score at Week 12 | Baseline, Week 12
  The GUPI assesses the degree of symptoms in both men and women with genitourinary pain complaints over the last week, including experience of pain or discomfort in various areas, frequency of pain/discomfort, average pain/discomfort, frequency of urinary symptoms, and quality of life (QoL) impact
Frequency of Treatment-emergent adverse events (TEAEs) occurring in ≥2% of subjects | Baseline, Week 12
  Frequency of TEAEs occurring in ≥2% of subjects
Overall frequency of TEAEs by severity grade | Baseline, Week 12
  Overall frequency of TEAEs by severity grade

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ironwood Pharmaceuticals
Locations (53):
- United States (53):
  - Urology Associates of Mobile, Mobile, Alabama
  - Velocity Clinical Research, Mobile, Alabama
  - Ironwood Research Center, Scottsdale, Arizona
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Ironwood Research Center, Fresno, California
  - American Institute of Research, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - UCI Health, Orange, California
  - Ironwood Research Center, San Diego, California
  - Solano Regional Medical Group Sutter Regional Medical Foundation, Vacaville, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advanced Urology Institute-Daytona Beach, Daytona Beach, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Clinical Associates of Orlando, Orlando, Florida
  - Altus Research, Palm Springs, Florida
  - Precision Clinical Research, Sunrise, Florida
  - South Tampa Health Services, Tampa, Florida
  - Ironwood Research Center, Cartersville, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - First Urology PSC, Jeffersonville, Indiana
  - Clinical Associates Midwest, Overland Park, Kansas
  - Wichita Urology - Newton, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Ochsner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Bay State Clinical Trials, Watertown, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - Specialty Clinical Research of St. Louis-Objective Health, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Ironwood Research Center, Hackensack, New Jersey
  - New Mexico Clinical Research and Osteoporosis Center, Albuquerque, New Mexico
  - Urological Institute of Northeast New York, Albany, New York
  - Accumed Research Associates, Garden City, New York
  - The Arthur Smith Institute for Urology - New Hyde Park Location, New Hyde Park, New York
  - Columbia University Irving Medical Center, New York, New York
  - Ironwood Research Center, New York, New York
  - Atrium Health Wake Forest Baptist Medical Center - Urology, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Center for Pelvic Health and Urogynecology - Tower Health Medical Group, Reading, Pennsylvania
  - Ironwood Research Center, Charleston, South Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Houston Metro Urology, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Advances In Health Inc, Pearland, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - The Chronic Pelvic Pain Center, Vienna, Virginia
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Ironwood Pharmaceuticals, Inc. is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to deidentified/pseudonymized, individual, and trial-level data (analysis data sets), as well as other information (eg, protocols, statistical analysis plans, clinical study report synopses) for Phase 2 through 4 trials that are not part of an ongoing or planned regulatory submission or are from a terminated program.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: These clinical trial data can be requested by any qualified researchers who engages in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data user agreement. Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered. For more information on the process, or to submit a request, visit the link below.
URL: http://ironwoodpharma.com/responsibility/patients-research/